CLINICAL TRIAL: NCT00640731
Title: Study of the OmniWave Endovascular System in Subjects With Lower and Upper Extremity Deep Vein Thrombosis - SONIC I Study
Brief Title: Safety and Efficacy Study of OmniWave Endovascular System to Treat Deep Vein Thrombosis
Acronym: SONIC I
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: OmniSonics Medical Technologies, Inc. (Other)
Responsible Party: Melina Salerno, Senior Clinical Project Manager, OmniSonics Medical Technologies, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-US-001
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2008-03

CONDITIONS: Deep Vein Thrombosis
Keywords: DVT; Peripheral Vascular Disease; Venous Thrombosis; Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: OmniWave Endovascular System — Treatment with mechanical thrombolysis/thrombectomy

SUMMARY:
This is a prospective, multi-center single arm registry to assess the use of the OmniWave Endovascular System in subjects presenting with either lower or upper extremity acute (symptoms have been present for greater than or equal to 14 days) DVT.

ELIGIBILITY:
Inclusion Criteria:

* DVT confirmed by venographic and ultrasound imaging, which has been symptomatic for a maximum of 14 days, or diagnosed within past 14 days defined as either first episode (no prior history in affected segment), or recurrent episode.
* Written informed consent
* Agreement to comply with follow up requirements

Exclusion Criteria:

* Known R-L shunt, pulmonary A-V malformation
* Excessive tortuosity and/or sharp angulation in target treatment zone
* Isolated calf vein thrombosis
* Isolated DVT in veins peripheral to axillary vein
* Thrombus in peripheral vessel smaller than 5 mm
* Target treatment zone cannot be adequately accessed within the 100 cm working length of device

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-07 (Estimated); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Procedural success rate defined as at least 50% reduction in thrombus burden in each target treatment zone following use of the OmniWave Endovascular System | Post-Index procedure

SECONDARY OUTCOMES:
Death, clinically detectable PE, significant vessel damage in target treatment area | through 6 months post-index procedure
Restoration and maintenance of antegrade in-line flow in target treatment area | through 6 months post-index procedure
QOL SF-36 | through 6 months post-index procedure
Incidence of clinically significant hemolysis | Prior to discharge

CONTACTS AND LOCATIONS:
Overall Officials: John Aruny, MD, Principal Investigator — Yale University